CLINICAL TRIAL: NCT06792383
Title: Psychological and Psychiatric Assessment in Patients Eligible for Epilepsy Surgery
Acronym: PsychoSurgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PsychoSurgery
Record Dates: First submitted 2025-01-08; First posted 2025-01-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Focal Epilepsy With and Without Secondary Generalization
Keywords: epilepsy; quality of life; psychiatric symptoms; stigma
MeSH Terms: conditions — Epilepsy; Social Stigma

STUDY DESIGN:
Intervention Model Description: The following assessment tools will be proposed to patients:
  * Quality of Life in Epilepsy (QOLIE-31)26
  * • Dissociative Experience Scale (DES)27
  * • Symptom Checklist-90 (SCL-90)28
  * • Irritability Questionnaire (I-EPI)29
  * • Beck Depression Inventory II (BDI-II)30
  * • State-Trait Anxiety Inventory Y-1 e Y-2 (STAI)31
  * • Epilepsy Stigma Scale modificata32 These assessment tools are validated and used universally, and will allow the collection of information on the psychological and psychiatric functioning of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with drug-resistant focal epilepsy (Experimental): patients with drug-resistant focal epilepsy eligible for epilepsy surgery who will undergo the procedure immediately.
  Interventions: Diagnostic Test: quality of life

INTERVENTIONS:
Diagnostic Test: quality of life — The following assessment tools will be proposed to patients:
  * Quality of Life in Epilepsy (QOLIE-31)26
  * Dissociative Experience Scale (DES)27
  * Symptom Checklist-90 (SCL-90)28
  * Irritability Questionnaire (I-EPI)29
  * Beck Depression Inventory II (BDI-II)30
  * State-Trait Anxiety Inventory Y-1 e Y-2 (STAI)31
  * Epilepsy Stigma Scale modificata32 These assessment tools are validated and used universally, and will allow the collection of information on the psychological and psychiatric functioning of the patients.
  Other Names: psychiatric symptoms

SUMMARY:
The aim of the study is to describe the socio-demographic, clinical, psychological, and psychiatric characteristics of patients with drug-resistant focal epilepsy eligible for epilepsy surgery and any changes in these parameters over time after surgery. Additionally, the study seeks to describe the levels of quality of life, dissociative experiences, prevalence of various psychiatric symptoms, irritability, depressive symptoms, anxiety symptoms, and stigma perception in patients with drug-resistant focal epilepsy eligible for epilepsy surgery and any changes over time after surgery.

DETAILED DESCRIPTION:
The aim of the study is to describe the socio-demographic, clinical, psychological, and psychiatric characteristics of patients with drug-resistant focal epilepsy eligible for epilepsy surgery and any changes in these parameters over time after surgery. Additionally, the study seeks to describe the levels of quality of life, dissociative experiences, prevalence of various psychiatric symptoms, irritability, depressive symptoms, anxiety symptoms, and stigma perception in patients with drug-resistant focal epilepsy eligible for epilepsy surgery and any changes over time after surgery.

This longitudinal, non-pharmacological interventional clinical study will be conducted at the Clinical and Experimental Epileptology Unit of the Institute. The enrollment will last for 24 months, during which approximately 30 patients with drug-resistant focal epilepsy eligible for epilepsy surgery will be enrolled, from both genders, aged at least 18 years.

Two groups of patients eligible for epilepsy surgery will be enrolled:

* Study group: patients with drug-resistant focal epilepsy eligible for epilepsy surgery who will undergo the procedure immediately.
* Control group: patients with drug-resistant focal epilepsy eligible for epilepsy surgery who, due to the need for further investigations and evaluations, will undergo the surgery at least 1 year after the baseline.

For the study group, data will be collected at three time points:

* At the time of pre-surgical hospitalization (baseline)
* 6 months after epilepsy surgery, during the first post-surgical follow-up visit (FU1)
* 12 months after epilepsy surgery, during the second post-surgical follow-up visit (FU2)

For the control group, data will be collected at three time points as well:

* At the time of surgical indication (baseline)
* 6 months after baseline and before epilepsy surgery (FU1)
* 12 months after baseline and before epilepsy surgery (FU2) At all three data collection time points, clinical psychological interviews and the administration of questionnaires evaluating the study variables will be conducted for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older at the time of enrollment;
* Patients with drug-resistant focal epilepsy followed at the Institute for at least 6 months;
* Patients with drug-resistant focal epilepsy eligible for epilepsy surgery;
* Patients capable of providing informed consent to participate in the study and for the processing of personal data.

Exclusion Criteria:

* Patients with evident and/or diagnosed cognitive or psychiatric disorders that prevent participation in an interview, proper understanding of informed consent, or completion of questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Psychological characteristics | 6 years
  Description of the time course of the clinical, psychological, and psychiatric characteristics of patients with drug-resistant focal epilepsy eligible for epilepsy surgery

SECONDARY OUTCOMES:
Levels of quality of life | 6 years
  Description of the time course of the levels of quality of life, dissociative experiences, prevalence of various psychiatric symptoms, levels of irritability, depressive symptoms, anxiety symptoms, and stigma perception in patients with drug-resistant focal epilepsy eligible for immediate epilepsy surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marco de Curtis, MD, Principal Investigator — Clinical and Experimental Epileptology Unit, Fondazione IRCCS Istituto Neurologico Carlo Besta, Via G. Celoria 11, 20133 Milano, Italy
Locations (1):
- Foundation IRCCS Carlo Besta Neurological Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawant N, Ravat S, Muzumdar D, Shah U. Is psychiatric assessment essential for better epilepsy surgery outcomes? Int J Surg. 2016 Dec;36(Pt B):460-465. doi: 10.1016/j.ijsu.2015.06.025. Epub 2015 Jun 12. PMID 26079497
- [Background] Locharernkul C, Kanchanatawan B, Bunyaratavej K, Srikijvilaikul T, Deesudchit T, Tepmongkol S, Lertlum S, Tuchinda L, Shoungshotti C, Ounpak P. Quality of life after successful epilepsy surgery: evaluation by occupational achievement and income acquisition. J Med Assoc Thai. 2005 Sep;88 Suppl 4:S207-13. PMID 16623030
- [Background] Devinsky O, Penry JK. Quality of life in epilepsy: the clinician's view. Epilepsia. 1993;34 Suppl 4:S4-7. doi: 10.1111/j.1528-1157.1993.tb05916.x. PMID 8348904
- [Background] Deleo F, Quintas R, Pastori C, Pappalardo I, Didato G, Di Giacomo R, de Curtis M, Villani F. Quality of life, psychiatric symptoms, and stigma perception in three groups of persons with epilepsy. Epilepsy Behav. 2020 Sep;110:107170. doi: 10.1016/j.yebeh.2020.107170. Epub 2020 Jun 5. PMID 32512366
- [Background] Shneker BF, Fountain NB. Epilepsy. Dis Mon. 2003 Jul;49(7):426-78. doi: 10.1016/s0011-5029(03)00065-8. PMID 12838266
- [Background] Langfitt JT, Westerveld M, Hamberger MJ, Walczak TS, Cicchetti DV, Berg AT, Vickrey BG, Barr WB, Sperling MR, Masur D, Spencer SS. Worsening of quality of life after epilepsy surgery: effect of seizures and memory decline. Neurology. 2007 Jun 5;68(23):1988-94. doi: 10.1212/01.wnl.0000264000.11511.30. PMID 17548548
- [Background] Spencer SS, Berg AT, Vickrey BG, Sperling MR, Bazil CW, Haut S, Langfitt JT, Walczak TS, Devinsky O; Multicenter Study of Epilepsy Surgery. Health-related quality of life over time since resective epilepsy surgery. Ann Neurol. 2007 Oct;62(4):327-34. doi: 10.1002/ana.21131. PMID 17567854
- [Background] Tellez-Zenteno JF, Patten SB, Jette N, Williams J, Wiebe S. Psychiatric comorbidity in epilepsy: a population-based analysis. Epilepsia. 2007 Dec;48(12):2336-44. doi: 10.1111/j.1528-1167.2007.01222.x. Epub 2007 Jul 28. PMID 17662062
- [Background] Luoni C, Bisulli F, Canevini MP, De Sarro G, Fattore C, Galimberti CA, Gatti G, La Neve A, Muscas G, Specchio LM, Striano S, Perucca E; SOPHIE Study Group. Determinants of health-related quality of life in pharmacoresistant epilepsy: results from a large multicenter study of consecutively enrolled patients using validated quantitative assessments. Epilepsia. 2011 Dec;52(12):2181-91. doi: 10.1111/j.1528-1167.2011.03325.x. PMID 22136077